CLINICAL TRIAL: NCT01428167
Title: Is There Any Association Between Thyroid Cancer and Hashimotos Thyroiditis?
Brief Title: Hashimotos Thyroiditis and Thyroid Cancer
Acronym: Thyroid Cancer
Status: Completed | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 11-112
Record Dates: First submitted 2011-08-10; First posted 2011-09-02 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-06

CONDITIONS: Thyroid Cancer; Hashimotos Thyroiditis
Keywords: Thyroid cancer; Hashimotos thyroiditis; Thyroidectomy; Anti-inflammatory factors
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples with be stored to measure anti inflammatory factors.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Thyroidectomy: All patients undergoing thyroidectomy for a variety of indications.

SUMMARY:
Thyroid cancer (TC) is the most common endocrine malignancy. The association between inflammation and cancer is well established but the association between thyroiditis (inflammation of thyroid gland) especially Hashimoto's thyroiditis (HT) and thyroid cancer remains controversial. Chronic inflammation leads to a repeated cycle of cellular damage and subsequent healing which contributes to inappropriate cell proliferation and subsequent neoplastic transformation. One of the most common forms of Thyroiditis is Hashimoto's thyroiditis which is a chronic autoimmune inflammatory disease affects almost 5% of the population and is more common in women. For the first time, Dailey and Lindsay reported in 1955 an increased association between Hashimoto's Thyroiditis (HT) and thyroid cancer. They reported 35 thyroid cancers in 278 patients with Hashimoto's Thyroiditis, a prevalence of 17.7% which they considered higher than the general population . Since then, various studies have been done, some studies have reported an increased risk of malignancy in Hashimoto's thyroiditis; others have failed to find an association. Most of the studies that have been done to identify the association between Hashimoto's thyroiditis and thyroid cancer are retrospective. The purpose of this pilot case-control study is to identify the association of Hashimoto's thyroiditis and thyroid cancer, to determine if the presence of Hashimoto's thyroiditis has any affect on the complication of thyroidectomy and prognostic factors of thyroid cancer.

DETAILED DESCRIPTION:
AIM1: To identify the association between Hashimoto's Thyroiditis and thyroid cancer by comparing the prevalence of thyroid cancer in patients with Hashimoto's Thyroiditis and patients without Hashimoto's Thyroiditis who undergoing Thyroidectomy for a variety of indications in UTMB in 12 months period of the study.

AIM2: Compare Ultrasound (US) characteristics preoperatively in two groups of patients with thyroid cancer and Hashimoto's thyroiditis and patients with thyroid cancer but without Hashimoto's thyroiditis.

AIM3: compare prognostic factors including tumor diameter, vascular and capsular invasion, extra thyroid invasion, lymph node metastasis, distant metastasis in two groups of patients including patients with thyroid cancer and Hashimoto's thyroiditis and patients with thyroid cancer but without Hashimoto's thyroiditis.

AIM4: Compare the complication of surgery in patients with thyroid cancer and Hashimoto's Thyroiditis and patients with thyroid cancer but without Hashimoto's thyroiditis.

AIM5: Compare inflammatory factors in two group of patient with thyroid cancer and Hashimoto's Thyroiditis and patients with thyroid cancer but without Hashimoto's thyroiditis.

Coordinator in the ear, nose and throat (ENT) clinic will notify the assigned investigator about any patient admitted to UTMB for thyroidectomy. The investigator will meet and interview the patient to obtain the consent and fill out a data collection sheet which will include demographic data, history of thyroid disease, history of thyroid medications, history of radiotherapy of head and neck or radioactive iodine therapy, family history of thyroid disease or thyroid cancer. Patients meeting the inclusion criteria will be given the opportunity to participate in the study. All patients will have blood drawn. Blood samples will be stored in Endocrinology lab to measure Anti-TPO, Ca, PTH and inflammatory factors at the end of study. A chart review of all enrolled patients will be performed to obtain details of the preoperative thyroid U/S characteristics including echogenicity, texture, calcification, vascularity and TSH and Free T4 level. Postoperative histopathology evaluation will be done by a pathologist experienced in thyroid pathology. The diagnosis of Hashimoto's thyroiditis (HT ) will be made based on histopathology finding and AntiTPO level. The histopathology criteria for Hashimoto's thyroiditis (HT) must be seen in a normal region of the thyroid gland, distinct from the site of thyroid cancer. UTMB Subjects will be divided to two groups, subjects with Hashimoto's Thyroiditis and subjects without Hashimoto's Thyroiditis (control group).The prevalence of thyroid cancer will be compared in these two groups.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing thyroidectomy for a variety of indications at University of Texas Medical Branch in Galveston between June 2011-May 2012
* Age 18-80 years old

Exclusion Criteria:

History of previous radiotherapy to head and neck and History of radioactive iodine therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing thyroidectomy for a variety of indications at University of Texas Medical Branch in Galveston between June 2011-May 2012
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Number of Participants with thyroid cancer and Hashimoto's thyroiditis . | one year
  To identify the association between Hashimoto's Thyroiditis and thyroid cancer by comparing the prevalence of thyroid cancer in patients with Hashimoto's Thyroiditis and patients without Hashimoto's Thyroiditis who undergoing Thyroidectomy for a variety of indications in UTMB in 12 months period of the study.

SECONDARY OUTCOMES:
Thyroid Ultrasound characteristics in participants with thyroid cancer in the setting of thyroid inflammation. | one year
  Compare Ultrasound (US) characteristics preoperatively in two groups of patients with thyroid cancer and Hashimoto's thyroiditis and patients with thyroid cancer but without Hashimoto's thyroiditis.
Prognostic factors of thyroid cancer | one year
  compare prognostic factors including tumor diameter, vascular and capsular invasion, extra thyroid invasion, lymph node metastasis, distant metastasis in two groups of patients including patients with thyroid cancer and Hashimoto's thyroiditis and patients with thyroid cancer but without Hashimoto's thyroiditis.
Complication of thyroidectomy( Thyroid surgery) | 2 weeks
  Compare the complication of surgery in patients with thyroid cancer and Hashimoto's Thyroiditis and patients with thyroid cancer but without Hashimoto's thyroiditis.
Inflammatory factors level in Plasma sample | one year
  Compare inflammatory factors in two group of patient with thyroid cancer and Hashimoto's Thyroiditis and patients with thyroid cancer but without Hashimoto's thyroiditis.

CONTACTS AND LOCATIONS:
Overall Officials: LaDale St Clair, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston , Endocrine Department, Galveston, Texas, United States